CLINICAL TRIAL: NCT06324890
Title: PET-CT Imaging Features of Meibomian Glands
Status: Recruiting | Type: Observational
Sponsor: Zhongnan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 20240225
Record Dates: First submitted 2024-02-27; First posted 2024-03-22 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2024-02

CONDITIONS: MGD-Meibomian Gland Dysfunction; Positron-Emission Tomography; Dry Eye
MeSH Terms: conditions — Meibomian Gland Dysfunction; Dry Eye Syndromes

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Analysis the results of Dry eye analysis results and PET-CT imaging comprehensively

DETAILED DESCRIPTION:
Medical records of patients who visited the ophthalmology department between January 2021 and December 2023 and had a PET-CT examination in our hospital within one month were collected. The dry eye analysis results of all patients were collected, and the lacrimal river height, tear film rupture time and meibomian gland grade were counted. The results of PET-CT were collected and the SUV values of the tarsal gland were calculated.

ELIGIBILITY:
Inclusion Criteria:

* Patients who visited the ophthalmology Department of Zhongnan Hospital from January 2021 to December 2023 and had a PET-CT examination in the hospital within one month

Exclusion Criteria:

* Dry eye analysis was not performed
* History of eye surgery or trauma
* Other systemic diseases affecting the eyes

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients who visited the ophthalmology Department of Zhongnan Hospital from January 2021 to December 2023 and had a PET-CT examination in the hospital within one month
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-01-31 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Lacrimal river height | Within a month of the PET imaging
  Measured by dry eye analyzer machine
Tear break-up time | Within a month of the PET imaging
  Measured by dry eye analyzer machine
Tear-film lipid layer thickness | Within a month of the PET imaging
  Measured by dry eye analyzer machine
Meibomian glands two-dimensional digital infrared images | Within a month of the PET imaging
  Measured by dry eye analyzer machine

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongnan Hospital of Wuhan University, Wuhan, Hubei, China